

# JAWATANKUASA ETIKA PENYELIDIKAN (MANUSIA) – JEPeM USM UNIVERSITI SAINS MALAYSIA

# TEMPLATE BORANG MAKLUMAT DAN KEIZINAN PESERTA TEMPLATE OF PARTICIPANT INFORMATION SHEET AND CONSENT FORM

(PROJEK PENYELIDIKAN) (RESEARCH PROJECT) <u>CONTOH</u> <u>ATTACHMENT B</u>

## RESEARCH INFORMATION

Research Title: A structural equation model and effects of music on mental, mindfulness,

psychological skills and sports performance among young basketball

players in Shandong Province, China

Name of main Researcher: SHUAI YING

Name of main supervisor: DR. KUEH YEE CHENG

Name of co-supervisor: ASSOC. PROF. DR. GARRY KUAN PEI ERN, ASSOC. PROF. DR. NAJIB MAJDI

**BIN YAACOB** 

#### INTRODUCTION

Your child (15 to 17 years) and you (parent/guardian) are invited to take part voluntarily in a cross-sectional research. This research is entitled A structural equation model and effects of music on mental, mindfulness, psychological skills and sports performance among young basketball players in Shandong Province, China. It is important to read and understand the research information before agreeing to allow your child to participate in this research study. If you agree to participate, you will receive a copy of this form to keep for your records or future reference. There will be 625 students, aged 15-17 years old participating in this study.

For study 1, <u>This study requires participants to complete the questionnaire and will take approximately</u> 30 minutes to complete. About 625 high school students from 1,2,3 grades will participate in the study. The validation process of the questionnaires will be translated using the Brislin method, with forward and backward translation.

For study 2, we will develop a music intervention program which is suitable for young basketball players in Shandong Province, China. This study will require participants to complete questionnaires and music intervention for basketball training. This study examine effects of music exercise on mental and sports performance of change among youth basketball players in China. 39 physically healthy athletes, age range between 15 to 17 years old will be recruited for this study. All participants will then be randomly assigned into 3 intervention groups and undergo 8 weeks (12 sessions) of the intervention period. The 3 intervention groups are: (i) general music intervention group; (ii) preferred music intervention group; and (iii) no music. Questionnaires and sports performance tests will be administered during the intervention.

#### **PURPOSE OF THE STUDY**

The purpose of this research is to examine the relationship between mental energy, mental toughness, mindful attention awareness, psychological skills and sport performance, as well as the effect of music exercise on mental and sports performance of change among youth basketball players in China.

#### **PARTICIPANTS CRITERIA**

The research team members will discuss your child's eligibility to participate in this study. It is important that you are completely truthful with the researcher including your child's health history.

For Study 1:The Inclusion Criteria includes: Youth basketball players with China nationality. Youth basketball players aged 15-17 years old. Youth basketball players who are understand the information that explained by the researcher and agree to be included in the study.

Exclusion Criteria includes: Youth basketball players that have any mental disorders (identified by the teachers). Your child should not participate in this study if he/she doesnot meet all the qualification stated above.

For Study 2:The Inclusion Criteria includes: Youth basketball players with China nationality. Youth basketball players aged 15-17 years old. Youth basketball players who are able to fulfil the given questionnaires before and after the intervention given. The athletes were members of the same team and had the same weekly training frequency, diet and routine before and after the intervention.

Youth basketball players had at least 2 years of training experience, no recent competition commitments, statistically insignificant differences in height and weight and BMI.

Exclusion criteria includes:Youth basketball players who unwilling to participate in the intervention phase.Youth basketball players with disabilities that avoiding them from being physically active. **Potential** medical problems that compromised participation or performance in the study

Withdrawal criteria: Participants are free to redraw from the study at any time without any penalty or disadvantage in the school.

You should not participate in this study if you do not meet all the qualification above or if you remember filling this questionnaire recently.

#### STUDY PROCEDURES

Promotional poster will be published throughout the entire club on theirvoluntary to participate as a participant. A brief description will be conductedfor those interested involve with the study.

If you agree to participate in this study, you will be asked to answerquestionnaires which consists of several sections: (1)Mental energy, (2)mental toughness, (3)psychological skills, and (4)mindfulness. The survey would take about 30 - 40minutes to complete.

Students who are injured ordo not want to participate in this study were excluded from the study. The Transtheoretical Model Questionnaire and the Social-ecological Questionnaire, inform consent and participant demographic sheet withinclusion and exclusion criteria will be distributed and filled by the subjects before further participation.

This is a pre-test – intervention – post-test design. In the pre-test, participants firstly completed a demographic questionnaire. Next, they completed the mood scale before and after competing in a simulated competition as appropriate. Participants were then randomly assigned into three interventions research conditions (i) with music intervention group; (ii) without music intervention group; and (iii) with a preference for the music intervention group. Participants then undertook 12 sessions of training with or without music over eight weeks. Following the eight weeks of training, a post-test in a simulated competition will be conducted under equivalent conditions to the pre-test.

Participants completed the mental energy, mental toughness, mindful attention awareness, psychological skills, mood, arousal, feelings, before and after the simulated competition. Psycho-physiological indicators of Sports performance. After post-testing, 9 participants (three in each condition) will be randomly selected to further explore the subjective experiences of the intervention (3 groups) using a short interview. The researcher will be involved throughout the study and will monitor the process every step of the way.

#### RISKS

There is no foreseen potential risk to the general students. The risk of music intervention is very minimum. To prevent the potential risk of moderate to intense exercise during the basketball for young people, we have trained physical education teachers with CPR certified who will be going to implement the intervention study and all participants had purchased their personal accident insurance (team regulation). In case of study related injury, the PE teachers will be bringing the participants for medical treatment

#### REPORTING HEALTH EXPERIENCES

Please contact, at any time, the following researcher if you experience any health problem either directly or indirectly related to this study.

Mr. SHUAI YING [P-UD0029/21(R)] at <contact No. +86 17606333635>

### **PARTICIPATION IN THE STUDY**

Your taking part in this study is entirely voluntary. You may refuse to take part in the study or you may stop your participation in the study at anytime, without any penalty or loss of benefits to which you are otherwise entitled. This study is unsponsored and all costs of the study are the responsibility of the researcher. Your participation also may be stopped by the research team without your consent if in any form you have violated the study eligibility criteria. The research team member will discussed with you if the matter arises.

### POSSIBLE BENEFITS [Benefit to Individual, Community, University]

Direct benefit - All participants will be having better lifestyles by performing music interventions. Besides, participants will not receive any insurance or compensation in the form of money but a certificate of appreciation from this study. There will no compensation for the participant or the participant'family or dependents in case of study-related injuries. This is because all participants had purchased their personal accident insurance (team regulation). Indirect benefit – The procedures of this study will be given to the students without cost. And schools and communities will become more aware of the benefits of music interventions exercise and become more involved. All participants will be able to obtain the research outputs through the research publication after the study has completed.

#### **QUESTIONS**

If you have any question about this study or your rights, please contact;

SHUAI YING SCHOOL OF MEDICAL SCIENCES USM Health Campus No. Tel: +86 17606333635

Email: cabe-wang@student.usm.my

Dr Kueh Yee Cheng School of Medical Sciences (PPSP) USM Health Campus No. 7el: 019-7666159

No. Tel: 019-7666159 Email: <a href="mailto:yckueh@usm.my">yckueh@usm.my</a>

Assoc. Prof. Dr Garry Kuan Pei Ern Exercise and Sports Science Unit School of Health Sciences (PPSK) USM Health Campus

No. Tel: 012-7228847 Email: garry@usm.my

If you have any questions regarding the Ethical Approval or any issue / problem related to this study, please contact:

Mr. Mohd Bazlan Hafidz Mukrim Secretary of Human Research Ethics Committee USM Division of Research & Innovation (R&I) USM Health Campus

Tel. No.: 09-767 2354 / 09-767 2362

Email: bazlan@usm.my

OR

Miss Nor Amira Khurshid Ahmed Secretariat of Human Research Ethics Committee USM Research Creativity & Management Office (RCMO) USM Main Campus, Penang

Tel. No.: 04-6536537 Email: noramira@usm.my

### CONFIDENTIALITY

Your information will be kept confidential by the researchers and will not be made publicly available unless disclosure is required by law.

Data obtained from this study that does not identify you individually will be published for knowledge purposes.

Your original records may be reviewed by the researcher, the Ethical Review Board for this study, and regulatory authorities for the purpose of verifying the study procedures and/or data. Questionnaires will be stored for at least 5 years with number coding. The questionnaire will not be open to the public. The study will not provide any feedback on the results. However, participants can obtained the study outcomes information through the study publication in future. There are no plan to develop this study into a commercial product and thus, the participant will not receive monetary or other benefit from such development. Your information may be held and processed on a computer. Only research team members are authorized to access your information.

By signing this consent form, you authorize the record review, information storage and data process described above.

#### **SIGNATURES**

To be entered into the study, you or a legal representative must sign and data the signature page [ATTACHMENT S or ATTACHMENT G (for genetic sample only) or ATTACHMENT P]

# Subject Information and Consent Form (Signature Page)

Research Title: A structural equation model and effects of music on mental, mindfulness,

psychological skills and sports performance among young basketball

players in Shandong Province, China

Researcher's Name: WANHG SHAOSHEN
Name of main supervisor: DR. KUEH YEE CHENG

Name of co-supervisor: ASSOC. PROF. DR. GARRY KUAN PEI ERN, ASSOC. PROF. DR. NAJIB

MAJDI BIN YAACOB

To become a part this study, you or your legal representative must sign this page. By signing this page, I am confirming the following:

- I have read all of the information in this Patient Information and Consent Form including any information regarding the risk in this study and I have had time to think about it.
- All of my questions have been answered to my satisfaction.
- I voluntarily agree to be part of this research study, to follow the study procedures, and to provide necessary information to the doctor, nurses, or other staff members, as requested.
- I may freely choose to stop being a part of this study at anytime.
- I have received a copy of this Participant Information and Consent Form to keep for myself.

| Participant Name | |
|-------------------------------------------------------|-----------------|
| Participant I.C No | |
| Signature of Participant or Legal Representative | Date (dd/MM/yy) |
| Name of Individual Conducting Consent Discussion | |
| Signature of Individual Conducting Consent Discussion | Date (dd/MM/yy) |
| Name & Signature of Witness | Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insuranc

# Participant's Material Publication Consent Form Signature Page

Research Title: A structural equation model and effects of music on mental, mindfulness,

psychological skills and sports performance among young basketball

players in Shandong Province, China

Researcher's Name: SHUAI YING

Name of main supervisor: DR. KUEH YEE CHENG

Name of co-supervisor: ASSOC. PROF. DR. GARRY KUAN PEI ERN, ASSOC. PROF. DR. NAJIB

MAJDI BIN YAACOB

To become a part this study, you or your legal representative must sign this page.

By signing this page, I am confirming the following:

- I understood that my name will not appear on the materials published and there have been efforts to make sure that the privacy of my name is kept confidential although the confidentiality is not completely guaranteed due to unexpected circumstances.
- I have read the materials or general description of what the material contains and reviewed all photographs and figures in which I am included that could be published.
- I have been offered the opportunity to read the manuscript and to see all materials in which I am included, but have waived my right to do so.
- All the published materials will be shared among the medical practitioners, scientists and journalist world wide.
- The materials will also be used in local publications, book publications and accessed by many local and international doctors world wide.
- I hereby agree and allow the materials to be used in other publications required by other publishers with these conditions:
- The materials will not be used as advertisement purposes nor as packaging materials.
- The materials will not be used out of contex i.e.: Sample pictures will not be used in an article which is unrelated subject to the picture.

| Participant Name | |
|-------------------------------|-----------------------------------------|
| <br>Participant I.C No. | Participant's Signature Date (dd/MM/yy) |
| <br>Name and Signature of Inc | dividual Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insurance.